CLINICAL TRIAL: NCT01165567
Title: Phase 4 Study of Sarpogrelate That Prevent Contrast-induced Nephropathy
Brief Title: The Prevention of Contrast Induced Nephropathy by Sarpogrelate in Patients With Chronic Kidney Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Boramae Hospital (Other)
Responsible Party: Seoul National University Boramae Hospital, Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20091104/06-2009-123/89
Record Dates: First submitted 2010-07-19; First posted 2010-07-20 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — sarpogrelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sarpogrelate 300 mg per day (Experimental): Patients in the sarpogrelate group receive sarpogrelate 300 mg per day for 24 hours before exposure to contrast agent.
  Interventions: Drug: sarpogrelate
- No sarpogrelate medication (No Intervention)

INTERVENTIONS:
Drug: sarpogrelate — sarpogrelate, 300mg/day,duration: 4 weeks
  Other Names: Anplag
  Arms: sarpogrelate 300 mg per day

SUMMARY:
Background:

Contrast-induced nephropathy (CIN) is a serious clinical problem associated with increased morbidity and mortality, particularly in patients with chronic renal insufficiency. Although some agents including hydration with saline are being prescribed to prevent renal deterioration in these high risk patients, their efficacy is not clear defined and debatable. Therefore additional prophylactic pretreatments are needed.

Methods/Design:

Present study aims to investigate differences in occurrence of CIN after sarpogrelate premedication in patients with chronic kidney disease (CKD). 268 participants, aged 20-85 years with a clinical diagnosis of CKD will be recruited. They will be randomly allocated to one of two conditions: (i) a routine treatment without sarpogrelate group (ii) routine treatment with sarpogrelate (a fixed-flexible dose of 300 mg/day). The primary outcome is the occurrence of CIN during 4 weeks after receiving contrast agent.

Discussion:

As of May 2010, there were no registered trials evaluating the therapeutic potentials of sarpogrelate in preventing for CIN. If sarpogrelate decreases the worsening of renal function and occurrence of CIN, it will provide a safe, easy and inexpensive treatment option.

DETAILED DESCRIPTION:
All patients with CKD scheduled for CAG will be eligible, assuming their ability to understand the character and individual consequences of participation as well as giving written informed consent. CKD is defined as estimated glomerular filtration rate (eGFR) <60 mL/min per 1.73 m2 using modification of diet in renal disease (MDRD) formula or serum creatinine (Cr) > 1.5 mg/dL.

The MDRD formula was defined in the following way. Where the Cr concentration is in mg/dL:

eGFR = 186 × serum Cr-1.154 × Age-0.203 × (0.742 if female) Exclusion criteria are age less than 20 years or more than 85 years, liver cirrhosis greater than or equal to Child class B, decreased serum platelet level (< 100,000/uL), patients who received or are schedule to receive percutaneous renal intervention, currently are taking anticoagulation drugs, unable to give informed consent. Patients in shock, maintaining hemodialysis, hemofiltration, peritoneal dialysis will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* patient with chronic kidney disease scheduled for coronary angiogram

Exclusion Criteria:

* age less than 20 years or more than 85 years
* liver cirrhosis greater than or equal to Child class B
* decreased serum platelet level (< 100,000/uL)
* patients who received or are schedule to receive percutaneous renal intervention
* currently are taking anticoagulation drugs
* unable to give informed consent

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
incidence of contrast-induced nephropathy | within 48 hours after using a contrast agent
  The primary outcome of the study is the incidence of CIN, defined as either a greater than 25 percent increase of serum Cr or an absolute increase in serum Cr of 0.5 mg/dL within 48 hours after using a contrast agent

SECONDARY OUTCOMES:
occurrence of CIN | at 4 weeks after using a contrast agent
  Clinical endpoint measurements are conducted in-hospital and at 4 weeks. Cr concentration is measured at admission, every day for the next two days after contrast exposure, and at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Ki YJ, Kwon SA, Kim HL, Seo JB, Chung WY. The Prevention of Contrast Induced Nephropathy by Sarpogrelate: a Prospective Randomized Controlled Clinical Trial. J Korean Med Sci. 2019 Oct 21;34(40):e261. doi: 10.3346/jkms.2019.34.e261. PMID 31625293
- [Derived] Park K, Chung WY, Seo JB, Kim SH, Zo JH, Kim MA, Park YB. The prevention of contrast induced nephropathy by sarpogrelate in patients with chronic kidney disease: a study protocol for a prospective randomized controlled clinical trial. Trials. 2010 Dec 20;11:122. doi: 10.1186/1745-6215-11-122. PMID 21167080